CLINICAL TRIAL: NCT06773936
Title: A Phase II Trial of Asciminib, Dasatinib, Prednisone, and Blinatumomab for Participants With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia
Brief Title: Adding Asciminib to Usual Treatment for Adults With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21CTP.LEUK01; CABL001AUS11R (Other: Novartis)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia; CD19+ Acute Leukemia
Keywords: PH+ALL; ALL; Philadelphia Chromosome Positive; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Induction Phase — Asciminib, Dasatinib, Prednisone, and Methotrexate
Drug: Re-Induction Phase — Blinatumomab, Dasatinib, Methotrexate, and Dexamethasone
Drug: Post-Remission — Blinatumomab, Dasatinib, Methotrexate and Dexamethasone
Drug: Maintenance — Asciminib, Dasatinib, Prednisone, and Methotrexate

SUMMARY:
This phase II trial is to answer the question of "can adding the study drug, asciminib to usual treatment improve how chemotherapy works against Ph+ Acute Lymphoblastic Leukemia (ALL) and is this approach better than the usual approach for Ph+ALL?"

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of major molecular remission (MMR) by polymerase chain reaction (PCR) for BCR-ABL at day 85 in newly diagnosed participants with Philadelphia-chromosome positive Ph+ acute lymphoblastic leukemia (ALL) treated with asciminib, dasatinib and prednisone.

SECONDARY OBJECTIVES:

I. To estimate the rate of complete remission (with and without complete count recovery, CR/CRi) at day 85 in this participant population.

II. To describe disease-free survival (DFS) in this participant population. III. To estimate overall survival (OS) in this participant population. IV. To estimate the frequency and severity of toxicities in this participant population.

V. To estimate the rate of measurable residual disease remission by flow cytometry (MRD Flow) at day 85 in this participant population.

VI. To compare rates of MMR by PCR and MRD flow remission in this participant population.

VII. Among participants who achieve MMR, to estimate the cumulative incidence of relapse from MMR in this participant population.

VIII. To describe attainment and failure of MR3.0, MR4.0 and MR4.5 at day 85 in this participant population.

IX. To estimate the rate of complete remission with undetectable MRD levels by flow cytometry (MRDundetectable CR) in this participant population.

X. To estimate duration of MMR in this participant population. XI. To estimate duration of MR4.0 in this participant population. XII. To estimate time to treatment failure in this participant population. XIII. To describe event-free survival (EFS) in this participant population.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate and describe the genes and pathways associated with response (molecular response) to therapy.

II. To describe the spectrum of mutations observed, and the timing of their emergence, in resistant/relapse samples.

III. To bank specimens for future correlative studies.

OUTLINE: Patients will have their phase of treatment determined by their responses tested by blood and bone marrow tests.

PHASE 1 TREATMENT (INDUCTION):

Phase 1 treatment may last up to 12 weeks. Patients will start with 4 weeks of treatment. Patients will receive Asciminib every day with a combination of other drugs. After 4 weeks of Phase 1 treatment, patients will be testing to see how the leukemia is responding. If There are no more signs of leukemia, the patients will receive 8 more weeks of Phase 1 treatment. if there are still signs of leukemia, patients will receive 4 more weeks of Phase 1 treatment and then will be tested again. If there are no signs of leukemia, they will receive 4 more weeks of Phase 1 treatment for a total of 12 weeks. If there are no signs of leukemia, patients will start Phase 2 treatment. If there are still signs of leukemia, the patients will start Re-induction treatment. Re-Induction treatment may last up to 12 weeks. Patients will start with 6 weeks of treatment. Patients will receive Blinatumomab every day for 28 days and Dasatinib every day for 42 days. After weeks of treatment, patients are tested and if there are no signs of leukemia, patients will start Phase 2 treatment. If there are still signs of leukemia, patients will repeat 6 weeks of Re-induction treatment. After repeating 6 weeks of Re-induction treatment if there are no signs of leukemia, patients will start Phase 2 treatment. If there are still signs of leukemia, patients will stop treatment in the study.

PHASE 2 TREATMENT (POST-REMISSION):

Phase 2 treatment will last up to 18 weeks. Patients will receive treatment in cycles of 42 days. There are 3 cycles of Phase 2 treatment. Patients will receive Blinatumomab every day for days 1-28 of each cycle and Dasatinib every day of each cycle. After Phase 2 treatment, patients will be tested. If there are no signs of leukemia, patients will start Phase 3 treatment. If there are signs of leukemia, patients will stop treatment in the study.

PHASE 3 TREATMENT (MAINTENANCE):

Patients will receive maintenance treatment for as long as it helps them. Phase 3 Treatment is given in 28-day cycles. Patients will receive Asciminib every day of each cycle, for up to five years from the time they started the study. Patients will take Dastinib every day of each cycle for as long as it helps them and Prednisone days 1-5 of each cycle for 18 cycles. Patients will stop treatment if the leukemia comes back or if side effects become too severe.

After completion of study treatment, patients are followed up on every 3 months for the first two years, and every 6 months until five years after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a new diagnosis of Philadelphia chromosome positive (Ph+) ALL by cytogenetics, FISH, or polymerase chain reaction (PCR). Diagnostic specimens must be submitted to the site's local CLIA-approved cytogenetics laboratory and results (cytogenetics, FISH, or PCR) must confirm Ph status prior to registration.
* Participants must have BCR-ABL status (p190 or p210) performed but results don't need to be back prior to Step 1 registration.
* Participants must have evidence of CD19+ ALL in their marrow or peripheral blood with at least 20% lymphoblasts present in blood or bone marrow collected within 28 days prior to registration. Immunophenotyping of the blood or marrow lymphoblasts must be performed to determine lineage. Appropriate marker studies including CD19 (B cell) must be performed. If a bone marrow aspirate cannot be obtained despite an attempt (dry tap), appropriate Immunohistochemistry (IHC) testing, including CD19, must be performed on the bone marrow biopsy to determine lineage. Participants with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible. CD19+ is defined as > 20% expression by flow cytometry or IHC.
* Participants must have recovered from any prior major surgery adverse effects within 14 days prior to registration, to the satisfaction of the local investigator.
* Participants must be ≥ 60 years old, or, if participants are under 60 years of age, they are not suitable for standard intensive induction chemotherapy at the discretion of the local investigator or must have refused standard intensive chemotherapy.
* Participants must have a lumbar puncture to determine CNS involvement of ALL within 14 days prior to registration. Note that intrathecal methotrexate administered during the pre-study lumbar puncture may count as the first dose of intrathecal therapy required as part of the study.
* Participants must have completed medical history and physical exam within 28 days prior to registration.
* Participants must have Zubrod/ECOG Performance Status of 0-3.
* Participants with extramedullary disease at diagnosis must have an MRI or CT scan with contrast of chest, neck, abdomen, pelvis, or whole body to obtain baseline values within 28 days prior to registration.
* Participants must have adequate pancreatic and liver function within 14 days prior to registration
* Participants must have a calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault Formula. This specimen must have been drawn and processed within 14 days prior to registration.
* Participants must have adequate cardiac function.
* Participants must be able to take oral medications and comply with the oral regimen.
* Participants with history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration, if indicated.
* Participants with known history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants must have an undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration, if indicated.
* Participants must agree to have peripheral blood and bone marrow specimens submitted for translational studies.
* Participants must be offered the opportunity to participate in specimen. banking

Exclusion Criteria:

* Participants must not have known lymphoid blast crisis of CML or have received previous TKI therapy for their CML.
* Participants must not have received any prior chemotherapy, investigational agents, radiation therapy, or other therapy for the treatment of ALL other than the following for a maximum of 7 days: FDA-approved TKI therapy, steroids, hydroxyurea, leukapheresis, and intrathecal chemotherapy.
* Participants must not be receiving any immunosuppressive therapy.
* Participants must not have received a prior autologous or allogeneic hematopoietic stem cell transplant.
* Participants must not have received any monoclonal antibody therapy within 42 days prior to registration.
* Participants must not have a history or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, active ALL in the CNS confirmed by CSF analysis, or other significant CNS abnormalities.
* Participants must not have a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen (in the opinion of the treating physician).
* Participants must not have systemic fungal, bacterial, viral or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment) as determined by the local investigator.
* Participants must not have clinically significant pericardial effusion, ascites or pleural effusion based on chest CT or x-ray or echocardiogram within 28 days prior to registration. Exceptions: if the effusion is suspected to be related to leukemia, the participant may have pericardial effusion ≤ Grade 2 or pleural effusion ≤ Grade 1.
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 24 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen.
* Participants must not have clinically significant autoimmune disease.
* Participants must not be receiving any proton pump inhibitors at the time of registration.
* Participants must not have impairment of gastrointestinal function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome). Participants who have had a gastrectomy are eligible.
* Participants must not have a history of or current acute pancreatitis, chronic pancreatitis, or any ongoing pancreatic disease.
* Participant must not have uncontrolled intercurrent illness.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Major molecular remission by polymerase chain reaction for BCR-ABL | Up to 100 days after treatment start
  Major molecular remission (MMR), also known as MR3.0, is defined as BCR-ABL transcript levels (expressed as a percentage compared with the ABL control gene) ≤ 0.1% based on PCR at day 85.

SECONDARY OUTCOMES:
Rate of Complete Remission (with and without complete count recovery, CR/CRi) | Up to 100 days after treatment start
  Complete response rate is measured by the number of participants achieving complete remission (CR) or complete remission with incomplete platelet recovery (CRi) rate. CR is defined as having <5% marrow aspirate blasts, ANC >1,000/mcL, platelets > 100,000/mcL, no blasts in peripheral blood, and C1 extramedullary disease status. CRi is the same as CR but platelet count may be <= 100,000/mcL and/or ANC <=1,000/mcL.
Disease-free Survival | Up to 5 years.
  Measured from the date the participant first achieves CR or CRi until relapse from CR/CRi or death from any cause. Observations will be censored on the day of last contact for participants last known to be alive in CR/CRi.
Overall Survival | Up to 5 years
  From the day of Step 1 registration on study until death from any cause with observations censored on the day of last contact for participants last known to be alive.
Incidence of Adverse Events | Up to 5 years
  Number of participants with Grade 3-5 adverse events that are possibly, probably or definitely related to study drug are reported by given type of adverse event. Adverse Events are reported using CTCAE v 5.0.
Rate of Measurable Residual Disease Remission by Flow Cytometry (MRD Flow) | Up to 100 days after treatment start
  Measurable residual disease (MRD) remission is defined as undetectable MRD levels by flow cytometry.
Major molecular remission and measurable residual disease remission by flow cytometry | Up to 100 days after treatment start
  Comparison of rates of major molecular remission by polymerase chain reaction (MMR) and measurable residual disease remission by flow cytometry (MRD Flow).
Relapse from Major Molecular Remission (MMR) | Up to 5 years
  Cumulative incidence of relapse from MMR, defined as BCR-ABL transcript levels (expressed as a percentage compared with the ABL control gene) > 0.1% based on PCR.
Molecular Response 4.0 (MR4.0) Rate at Day 85 | Up to 100 days after treatment start
  MR4.0 is defined as a 4.0-log reduction, relative to baseline, of the BCR-ABL/ABL ratio based on PCR. This response is equivalent to a value of <= 0.01% when reported on the International Scale.
Molecular Response 4.5 Rate at Day 85 | Up to 100 days after treatment start
  MR4.5 is defined as a 4.5-log reduction, relative to baseline, of the BCR-ABL/ABL ratio based on PCR. This response is equivalent to a value of <= 0.0032% when reported on the International Scale.
Rate of Complete Remission with Undetectable MRD by Flow Cytometry | Up to 5 years
  Number of participants meeting criteria for complete remission (CR) and measurable residual disease flow remission (MRD Flow).
Duration of Major Molecular Remission by PCR | Up to 5 years
  Measured from the date the participant first achieves MMR until relapse from MMR or death from any cause. Observations will be censored on the day of last contact for participants last known to be alive in MMR.
Duration of MR4.0 by PCR | Up to 5 years
  Measured from the date the participant first achieves MR4.0 until relapse from MR4.0 or death from any cause. Observations will be censored on the day of last contact for participants last known to be alive in MR4.0.
Time to Treatment Failure | Up to 5 years
  From the day of Step 1 registration on study until treatment failure, or death due to any cause. Observations will be censored on the day of last contact for participants last known to be alive and failure free.
Event-free Survival | Up to 5 years.
  From the day of Step 1 registration on study until failure to achieve CR/CRi following induction or re-induction, relapse from CR/CRi, or death due to any cause. Observations will be censored on the day of last contact for participants last known to be alive in CR/CRi.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali S Advani, Principal Investigator — SWOG Network Cancer Center
Locations (2):
- United States (2):
  - University of Cincinnati Cancer Ctr-UC Medical Ctr, Cincinnati, Ohio
  - Baptist Memorial Health Care, Memphis, Tennessee